CLINICAL TRIAL: NCT03902171
Title: Outcomes Related to Use of Soberlink Within In-Home Addiction Treatment Program for Individuals With Alcohol Use Disorder
Brief Title: Soberlink Within In-Home Addiction Treatment Program
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: In-Home Addiction Treatment Institute, Inc. (Other)
Collaborators: Soberlink Healthcare LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SLIHAT-2019
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Primary diagnosis alcohol use disorder (AUD): Primary diagnosis of alcohol use disorder (AUD) population enrolled in In-Home Addiction Treatment Program.
  Interventions: Device: Soberlink
- Secondary diagnosis alcohol use disorder (AUD): Secondary diagnosis of alcohol use disorder (AUD) population enrolled in In-Home Addiction Treatment Program.
  Interventions: Device: Soberlink

INTERVENTIONS:
Device: Soberlink — Soberlink delivers real-time blood alcohol results to people who support individuals in recovery from alcohol use disorder. In-Home Addiction Treatment program Care Team monitors and responds to results as part of care to improve treatment outcomes.

SUMMARY:
The purpose of this study is to evaluate the impact of use of Soberlink on treatment experience for individuals with alcohol use disorder while enrolled in an In-Home Addiction Treatment program. Treatment engagement, feelings related to autonomy and empowerment, and overall quality of life will be evaluated. Although not the primary focus, recidivism and relapse will be measured.

DETAILED DESCRIPTION:
The study will include 30 Clients with a primary or secondary diagnosis of alcohol use disorder (AUD) and who are enrolled in Aware Recovery Care's In-Home Addiction Treatment program where Care Teams will monitor cloud-based breathalyzer results. Soberlink's cloud-based breathalyzer system will provide data to Care Team if the Client has relapsed or is not compliant with testing through the Soberlink System. Clients will use Soberlink for 180 days within context of routine alcohol use disorder treatment at Aware Recovery Care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between ages of 21-75 years old
* Subject active in In-Home Addiction Treatment Program (Aware Recovery Care)
* Subject admitted to program with American Society of Addiction Medicine (ASAM) Assessment score 1.5-2.5
* Primary or secondary diagnosis is alcohol use disorder
* Subject is willing to use Soberlink Device to provide Blood Alcohol Content (BAC)
* Subject is willing to discuss Soberlink test results with Care Team
* Subject is willing to sign Soberlink Client Agreement
* Subject is English speaking and reading

Exclusion Criteria:

* Alcohol use disorder is not a primary or secondary diagnosis
* Subject is not between ages of 21 and 75 years old
* Subject is currently taking anti-alcohol/craving medications (Antabuse, Campral, Vivitrol)
* Subject will not be in the United States through duration of study
* Subject is unwilling to properly use the device
* Subject is non-English speaking and reading
* Subject is a child, adolescent, cognitively impaired, diagnosed with a mental disorder involving depersonalization or active psychotic symptoms
* Active withdrawal/alcohol use within 72 hours of start of participation
* Subject is using Soberlink data for a child custody or legal consequence

Ages: 21 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects are active participants in Aware Recovery Care, an In-Home Addiction Treatment program with an active primary or secondary diagnosis of alcohol use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-09-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Retention in Treatment | 180 days duration of subject participation
  Participation in In-Home Addiction Treatment program using length of stay reports.
Brief Addiction Monitor questionnaire | Conducted monthly throughout 180 days duration of subject participation
  Measure change in client report of symptoms related to alcohol use disorder
Positive Outcomes Measures Survey | Completed at week 3 or 4 and Week 20 during 180 days duration of subject participation
  Measures changes in quality of life using client self-report inquiring about employment, connection to care team, community engagement using yes/no answer key
Client Survey Related to use of Soberlink | Completed at end of 180 days duration of subject participation
  Measures self-report of quality of life and experience with device using 5-point Likert scale (minimum Strongly Disagree, maximum Strongly Agree)

SECONDARY OUTCOMES:
Relapse Rates | Measured throughout 180 days duration of subject participation
  Occurrence of alcohol use
Compliance with Testing | Measured throughout 180 days duration of subject participation
  Occurrence of Missed Tests
Hospitalization | Measured throughout 180 days duration of subject participation
  Occurrence of Emergency Room and Inpatient hospital admissions
Detox and Residential Admissions | Measured throughout 180 days duration of subject participation
  Occurrence of residential treatment and detox admissions

CONTACTS AND LOCATIONS:
Overall Officials: Courtney MacNeill, LMSW, Principal Investigator — Research Associate
Locations (2):
- United States (2):
  - Aware Recovery Care, North Haven, Connecticut
  - Aware Recovery Care, Bedford, New Hampshire

IPD SHARING:
Plan to Share IPD: No